CLINICAL TRIAL: NCT06794125
Title: A Phase II/III Randomized Evaluation of Dose-escalation With Esophageal-sparing for Palliation of Intrathoracic Tumours (PREVENT)
Brief Title: An Evaluation of Dose-escalation for Intrathoracic Tumours
Acronym: PREVENT-LUNG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chris Goodman (Other)
Responsible Party: Sponsor-Investigator, Chris Goodman, MD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENT-LUNG
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancers
Keywords: lung cancer; radiation therapy; hypofractionated; esophageal-sparing; dose-escalated; intrathoracic
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Radiotherapy (Active Comparator): 20 Gray in 5 fractions or 30 Gray in 10 fractions.
  Interventions: Radiation: Radiation Therapy
- Experimental Radiotherapy (Experimental): 35 Gray in 5 fractions
  Interventions: Radiation: Hypofractionated Radiation Therapy

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Hypofractionated, dose-escalated, esophageal-sparing intensity modulated radiation therapy
  Arms: Experimental Radiotherapy
Radiation: Radiation Therapy — standard of care palliative thoracic radiotherapy using volumetric modulated arc therapy/intensity-modulating radiotherapy
  Arms: Standard Radiotherapy

SUMMARY:
This is a pragmatic trial with patients randomized between standard of care palliative thoracic radiation therapy (RT) vs. hypofractionated, dose-escalated, esophageal-sparing (HD-ES) intensity modulated radiation therapy (IMRT).

The investigators hypothesize that the use of advanced radiation planning techniques to optimize dose to esophagus will permit the safe delivery of a modestly dose-escalated five-fraction course of palliative radiation to intrathoracic malignancies. This approach aims to deliver higher biologically effective doses while improving toxicity when compared to conventional approaches with the goal of prolonging high-quality overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Intrathoracic tumour requiring palliative radiation, either for palliation of symptoms or prevention of progression that is expected to cause symptoms in the next 6 months (in the judgement of the enrolling investigator)
* Willingness and ability to provide informed consent
* Eastern Cooperative Oncology Group performance status 0-3
* Age 18 years or older
* Prior or planned systemic treatment (chemotherapy, immunotherapy, targeted agents) is permissible at the discretion of the treating medical oncologist
* Concurrent palliative radiotherapy to other metastatic sites is permissible at the discretion of the treating radiation oncologist.
* Life expectancy greater than 3 months

Exclusion Criteria:

* Prior thoracic radiotherapy which, in the opinion of the treating of radiation oncologist, precludes the delivery of further thoracic radiotherapy. If there has been prior thoracic radiotherapy, a composite of all RT plans must be created, and the dose constraints herein must still be met. An allowance for 10 percent repair is permitted if at least 12 months have passed between the prior radiotherapy and the trial protocol specified radiotherapy.
* Serious medical comorbidities which, in the opinion of the treating radiation oncologist, preclude the delivery of radiotherapy. This includes interstitial lung disease.
* Pregnant or lactating women
* Inability to attend the full course of radiotherapy or planned follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
time to definitive quality of life deterioration or death | from enrollment until 36 months post radiotherapy
  Defined as time from randomization to the first of:
  i. deterioration in Functional Assessment of Cancer Therapy: Lung Trial Outcome Index score by greater than or equal to 5 points compared to baseline score and with no subsequent improvement to within 5 points of baseline ii. death iii. last follow-up

SECONDARY OUTCOMES:
Quality of Life - Patient Reported Outcomes | From enrollment until 36 months post radiotherapy
  Measured via Functional Assessment of Cancer Therapy: Lung and EuroQol 5-dimension 5-level
Toxicity - Adverse Events that happen to a patient during the clinical trial | From enrollment until 36 months post radiotherapy
  Defined as incidence of Common Terminology Criteria for Adverse Events version 5 grade 2 and higher toxicity
Freedom from intrathoracic progression | From enrollment until 36 months post radiotherapy
  Defined as time from randomization to disease progression within the thorax, or last follow-up, whichever occurs first
Overall Survival | From enrollment until 36 months post radiotherapy
  Defined as time from randomization to death from any cause, or last follow-up, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - British Columbia Cancer Agency Center for the Southern Interior, Kelowna, British Columbia
  - London Health Sciences Center Research Institute (Formerly Lawson Research Institute), London, Ontario
  - Waterloo Regional Health Network, Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No